CLINICAL TRIAL: NCT01945632
Title: Effect of Root Planing on Surface Topography.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Juan Ignacio Rosales Leal, DDS, PhD., Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: root planing tophography
Record Dates: First submitted 2013-07-02; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- no treatment (No Intervention): Control group with no treatment.
- root planing (gracey curettes) (Experimental): treatment with root planing using conventional gracey curettes
  Interventions: Device: conventional gracey curettes
- Vertically oscillating ultrasonic device (Experimental): Treatment done with vertically oscillating ultrasonic device
  Interventions: Device: Vertically oscillating ultrasonic device
- Device: piezoelectric ultrasonic scraper (Experimental): Treatment using a piezoelectric ultrasonic scraper
  Interventions: Device: piezoelectric ultrasonic scraper

INTERVENTIONS:
Device: conventional gracey curettes
  Arms: root planing (gracey curettes)
Device: Vertically oscillating ultrasonic device
  Arms: Vertically oscillating ultrasonic device
Device: piezoelectric ultrasonic scraper
  Arms: Device: piezoelectric ultrasonic scraper

SUMMARY:
In a clinical trial of 19 patients, 44 single-rooted teeth will be randomly assigned to one of four groups for: 1) no treatment, 2) manual root planing with curettes; 3) root planing with piezoelectric ultrasonic scraper [PU]; or 4) root planing with vertically oscillating ultrasonic device [VOU]. Post-treatment, the teeth will be extracted and their topography analyzed in 124 observations with white light confocal microscopy, measuring the roughness parameters Rp, Rv, Rt, Ra, Rq, Rku, and Rsk.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing programmed tooth extraction for chronic advanced periodontitis.

Exclusion Criteria:

* Patients with no advanced periodontitis or patients that refused the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Surface roughness | two years

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, University of Granada, Granada, Granada, Spain